CLINICAL TRIAL: NCT05299632
Title: Pre-operative Localization of Parathyroid Adenomas Using F-18 PSMA PET/CT: A Pilot Study
Brief Title: F-18 PSMA for Localization of Parathyroid Adenoma
Status: Terminated | Type: Observational
Why Stopped: Interim results from the first three participants were not significant
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Raghuveer Halkar, Professor of Medicine: Radiology, Emory University
Other Study IDs: STUDY00003262
Record Dates: First submitted 2022-03-09; First posted 2022-03-29 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism | interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with biochemical and clinical evidence of primary hyperparathyroidism: Patients who have biochemical and clinical evidence of primary hyperparathyroidism and who are scheduled for routine surgery and preoperative imaging including 99mTc-MIBI planar imaging and SPECT/CT. Subjects who enroll in the study will receive one additional F-18PSMA PET/CT imaging study. F-18 PSMA imaging study will be scheduled on the same day as of the Tc-99m MIBI scan. Since F-18 PSMA PET/CT employs 511kEv annihilation photon, the lower energy if (140 KeV) of Tc-99m MIBI will not interfere.
  Interventions: Diagnostic Test: 99mTc-MIBI planar imaging and SPECT/CT.; Diagnostic Test: F- 18PSMA PET/CT imaging study

INTERVENTIONS:
Diagnostic Test: 99mTc-MIBI planar imaging and SPECT/CT. — Participants will undergo a Tc-MIBI scan and management will be as per the finding of the Tc MIBI scan which is the standard of care.
  Other Names: Standard of Care
Diagnostic Test: F- 18PSMA PET/CT imaging study — F-18 PSMA is an FDA-approved imaging agent used for PET/CT for evaluating metastatic prostate cancer. The findings of the images of F-18 PSMA will be shared with the referring /treating surgeon. However, the findings will not influence the management.
  Other Names: F- 18PSMA PET/CT

SUMMARY:
Parathyroid glands are in the neck and produce a substance called parathormone which maintains the calcium level in the blood. Sometimes one or more of the parathyroid glands become hyperactive and produce too much parathormone which causes increased calcium in the blood which can cause ill effects on multiple parts of the body.

Hyperactive glands are identified by Tc-99m Sestamibi (MIBI) scan which helps the surgeons to remove them with minimal risk to the patient. But about 30% of the time MIBI scan does not localize the hyperactive gland. There is some evidence that a new agent called F-18 PSMA (prostate-specific membrane antigen) can localize hyperactive parathyroid.

This study is being done to collect preliminary data to answer the question: Can imaging with the PET tracer, F-18 PSMA (Pylarify), prior to parathyroid surgery, provide better information to a surgeon than the standard of care imaging with MIBI scan? Patients who are scheduled for parathyroidectomy and are scheduled for imaging with MIBI scan prior to surgery will be asked to take part in this study.

This is a single institutional study to collect preliminary data to help do a larger study. Participants will get MIBI scan first, and the same day will get an F-18 PSMA scan which involves an injection in the vein, waiting an hour, and imaging of the neck and chest area for 10 minutes. The findings of F-18 PSMA will not interfere with the participant's management. Patients who participate will not directly benefit by participating in this study.

If the scanning method using F-18 PSMA shows better results than MIBI scan (standard of care) then the investigators will conduct a larger multi-institutional study. If the results prove that F-18 PSMA is better than the standard of care in the larger study, then patients with hyperactive parathyroid patients in the future will benefit.

DETAILED DESCRIPTION:
Hyperparathyroidism is an increasingly significant medical and public health condition in the United States. In the past two decades, the incidence of hyperparathyroidism has increased 300%, and currently, the disease affects at least 30,000 new patients each year in the United States. Parathyroid adenomas, parathyroid hyperplasia in primary and secondary hyperparathyroidism, and parathyroid carcinomas are increasing in frequency in this country. The causes of the increased incidence of hyperparathyroidism are not known. Multiple organs are affected in patients with hyperparathyroidism; notably, a worsening of the severity of osteoporosis, accelerated arteriosclerotic disease, and hypertension. Parathyroid carcinoma is no longer a rare illness, and there is no effective oncologic therapy for parathyroid carcinoma (which often is fatal).

Surgery is the only effective management for primary hyperparathyroidism. Preoperative localization of a parathyroid adenoma allows a unilateral neck exploration for the removal of the tumor. If localization is accurate, patients can undergo focal, minimally invasive parathyroidectomies with cure rates equivalent to conventional surgery, less anesthesia, improved cosmesis, and shorter hospital stays. Since this approach decreases both the duration of surgery and its morbidity, preoperative localization is gaining recognition as an important procedure. However, tumor localization can be challenging, in part because current imaging methodologies are sub-optimal, failing to identify the parathyroid tumor in as many as 30% of patients. In re-operative parathyroidectomy for persistent or recurrent hyperparathyroidism, localization plays an even greater role.

Unfortunately, current imaging modalities fail to localize 10-15% of tumors. Even though high-frequency ultrasound can detect parathyroid adenoma, the intra-operator variability and difficulties in patients with prior surgery often necessitate Tc-99m MIBI imaging which has become the standard of care for preoperative localization which allows minimally invasive surgery and decreases the surgical time. The most commonly used methodology uses dual-phase 99mTechnetium-sestamibi (99mTc-MIBI) scintigrams where images are acquired at 2 and 4 hours after radiopharmaceutical administration. Interference caused by the concentration of 99mTc-MIBI in the thyroid (in close proximity of parathyroid adenoma) is a major source of failure of localization. Even if sophisticated techniques such as SPECT/CT are used, the parathyroid tumor is not identified in as many as 30% of patients. Parathyroid glands are located very close to the thyroid and if a molecular probe concentrates in the thyroid as well as in the parathyroid then the thyroid background makes it difficult to localize parathyroid adenomas. Our preliminary data has shown that folate receptors are not expressed in thyroid tissue and thus folate receptor imaging becomes an innovative technique of imaging parathyroid pathologies without the interference from the signals from the thyroid. This proposal is based on our observations that human parathyroid tumor cells express high densities of folate receptors and thyroid cells do not. Prostate-specific membrane antigen (PSMA) labeled with Ga-68 PSMA has been in clinical use in Europe and Asia for more than 5 years. The FDA approved the F 18-labeled prostate-specific membrane antigen (PSMA)-targeted positron emission tomography (PET) imaging agent 18F-DCFPyL (Pylarify) for use in prostate cancer in May 2021. PSMA is also known as Glutamate carboxypeptidase II (GCP II), and N-acetyl-L-aspartyl-L-glutamate peptidase I (NAALADase I), NAAG peptidase. PSMA removes the g-linked glutamates from folate, providing deglutinated folate for absorption and nutrition and leaving single a-linked glutamate attached. The official gene name of PSMA is folate hydrolase 1 (FOLH1), reflecting its major role in folate uptake; however, PSMA usually acts as a glutamate carboxypeptidase (GCP), its major substrate can differ in different tissues. Yao et al. found that PSMA-expressing cells also demonstrated a 2-fold increased uptake of folate, suggesting that PSMA may be associated with folate transport. Ga-68 PSMA has been shown to concentrate in parathyroid adenoma and not in the thyroid (Pfob2019). Ga-68 has 68 minutes half-life, is generator produced, and is available for a few centers in California currently. F-18 PSMA had 120 minutes half-life and will be available as a unit dose. This makes F-18 PSMA an ideal agent for clinical use.

Researchers hypothesize that F-18 PSMA will give better pre-operative localization of parathyroid adenomas compared to the conventional imaging with 99mTc-MIBI. If this is the case the new method will provide more patients with a minimally invasive parathyroidectomy, reducing trauma to the patient and the healthcare costs. The project described here is designed to collect preliminary data for a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older.
* Patients will have biochemical and/or clinical evidence of primary hyperparathyroidism and be a surgical candidate for definitive parathyroid surgery.
* Ability to lie still for SPECT/CT and PET/CT scanning
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Age less than 18.
* Inability to lie still for SPECT/CT and PET/CT scanning.
* Cannot provide written informed consent.
* History of secondary hyperparathyroidism.
* Positive serum or urine pregnancy test within 24 hours of imaging

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have agreed for Tc-99m MBI parathyroid imaging and parathyroidectomy will be identified as potential participants
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Preoperative localization of the parathyroid adenoma by F-18-PSMA PET/CT | Up to 14 days after surgical removal of parathyroid adenoma
  Results of F-18 PSMA imaging regarding localization will be compared to surgical findings (Right: superior, inferior and/or Left: superior, inferior)
Preoperative size (mm) of the parathyroid adenoma by F-18-PSMA PET/CT | Up to 14 days after surgical removal of parathyroid adenoma
  Results of F-18 PSMA imaging will be compared to surgical findings described in the operative notes in the EMR
The sensitivity of the F-18-PSMA PET/CT uptake correlation with other pathologic criteria | Up to 14 days after surgical removal of parathyroid adenoma
  The lesion-based sensitivities of F-18-PSMA PET/CT uptake using surgical pathology of the parathyroid gland as the reference standard (The number of true positive image findings/The number of pathologically confirmed parathyroid adenoma or hyperplasia)
The specificity of the F-18-PSMA PET/CT uptake correlation with other pathologic criteria | Up to 14 days after surgical removal of parathyroid adenoma
  The lesion-based specificity of F-18-PSMA PET/CT uptake using surgical pathology of the parathyroid gland as the reference standard (The number of true negative image findings/The number of negative findings on surgical pathology)
The accuracies of the F-18-PSMA PET/CT uptake correlation with other pathologic criteria | Up to 14 days after surgical removal of parathyroid adenoma
  The lesion-based accuracy of the F-18-PSMA PET/CT uptake using surgical pathology of the parathyroid gland as reference standard (True positive and true negative image findings/The number of all surgical specimens)

CONTACTS AND LOCATIONS:
Overall Officials: Raghuveer Halkar, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory University Hospital (EUH), Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia

IPD SHARING:
Plan to Share IPD: No